CLINICAL TRIAL: NCT00150267
Title: A 5-Year Postmarketing Safety Study Of Xalcom In Patients With Open Angle Glaucoma Or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 912-OPT-0076-019
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2008-11-05 (Estimated); Status verified 2008-11

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Xalacom

INTERVENTIONS:
Drug: Xalacom

SUMMARY:
To estimate the frequency of patients with ocular/periorbital adverse events. To identify any possible long-term adverse consequences of increased iris pigmentation and to follow serious adverse events throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with open angle glaucoma and/or ocular hypertension requiring a reduction of IOP who were insufficiently responsive to topical betablockers

Exclusion Criteria:

* Previous and current treatment with any topical ophthalmic drug containing prostaglandins; any condition in which treatment with the betablocking agent, timolol, was contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 976 (Actual)
Dates: Start 2002-02

PRIMARY OUTCOMES:
Incidence of increase of iris pigmentation
incidence of development in darkening/lengthening/thickening of eyelashes and/or pigmentation of periorbital skin
occurrence of ocular/periorbital adverse events
occurrence of serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (72):
- Pfizer Investigational Site, Sydney, New South Wales, Australia
- Belgium (6):
  - Pfizer Investigational Site, Antwerp
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Edegem
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Liège
- Denmark (2):
  - Pfizer Investigational Site, København Ø
  - Pfizer Investigational Site, Odense C
- France (10):
  - Pfizer Investigational Site, Aire Sur Adour
  - Pfizer Investigational Site, Carcassonne
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Figeac
  - Pfizer Investigational Site, Haguenau
  - Pfizer Investigational Site, Le Cannet
  - Pfizer Investigational Site, Loos
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Versailles
- Germany (7):
  - Pfizer Investigational Site, Erlangen
  - Pfizer Investigational Site, Freising
  - Pfizer Investigational Site, Gerolzhofen
  - Pfizer Investigational Site, Hirschaid
  - Pfizer Investigational Site, Hösbach
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, Würzburg
- Greece (5):
  - Pfizer Investigational Site, Piraeus, Nikea-Piraeus
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Kavala
  - Pfizer Investigational Site, Pátrai
  - Pfizer Investigational Site, Thessaloniki
- Ireland (2):
  - Pfizer Investigational Site, Ennis, Co. Clare
  - Pfizer Investigational Site, Galway
- Italy (8):
  - Pfizer Investigational Site, Siena, Siena
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Perugia
  - Pfizer Investigational Site, Pisa
  - Pfizer Investigational Site, Torino
- Netherlands (3):
  - Pfizer Investigational Site, Alkmaar
  - Pfizer Investigational Site, Gouda
  - Pfizer Investigational Site, Rijswijk
- Spain (13):
  - Pfizer Investigational Site, Almería, Almeria
  - Pfizer Investigational Site, Palma de Mallorca, Balearic Islands
  - Pfizer Investigational Site, Badalona, Barcelona
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Terrassa, Barcelona
  - Pfizer Investigational Site, Lugo, Lugo
  - Pfizer Investigational Site, Getafe, Madrid
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Málaga, Malaga
  - Pfizer Investigational Site, Valencia, Valencia
  - Pfizer Investigational Site, Valladolid, Valladolid
  - Pfizer Investigational Site, Bilbao, Vizcaya
  - Pfizer Investigational Site, Zaragoza, Zaragoza
- Sweden (5):
  - Pfizer Investigational Site, Motala
  - Pfizer Investigational Site, Örebro
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Uppsala
  - Pfizer Investigational Site, Västerås
- United Kingdom (10):
  - Pfizer Investigational Site, Bristol, Gloucestershire
  - Pfizer Investigational Site, Cheltenham, Gloucestershire
  - Pfizer Investigational Site, Bolton, Lancs
  - Pfizer Investigational Site, Uxbridge, Middlesex
  - Pfizer Investigational Site, Norwich, Norfolk
  - Pfizer Investigational Site, Redhill, Surrey
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Lancaster
  - Pfizer Investigational Site, London

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=912-OPT-0076-019&StudyName=A%205-Year%20Postmarketing%20Safety%20Study%20Of%20Xalcom%20In%20Patients%20With%20Open%20Angle%20Glaucoma%20Or%20Ocular%20Hypertension